CLINICAL TRIAL: NCT06615414
Title: Clinical and Subclinical Cardiovascular Manifestations in Philadelphia Negative Myeloproliferative Neoplasms
Brief Title: Cardiovascular Manifestations in Ph-negative MPN
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Viola Waheed Saad, Assistant Lecturer, Assiut University
Other Study IDs: CVD in MPN
Record Dates: First submitted 2024-09-15; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Philadelphia Negative Myeloproliferative Neoplasms
Keywords: Cardiovascular manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 40 MPN patients: Inclusion criteria:
  * patients with confirmed diagnosis of myeloproliferative neoplasms of one of the following:
  * Essential thrombocythemia (ET)
  * Polycythemia vera (PV)
  * Primary myelofibrosis (PMF)
  * Adults aged 18 years and older.
  * who accept to participate in the study in Assiut university hospital.
  Exclusion criteria:
  * Patients with secondary erythrocytosis or thrombocytosis due to other underlying conditions (e.g., chronic hypoxia, tumors) will be excluded.
  * Patients who have experienced a myocardial infarction, stroke, heart failure, Hypertension, or significant cardiovascular event before diagnosis of MPN
  * Patients with severe comorbid conditions that could confound results, such as:
  * Severe renal or hepatic impairment
  * Active malignancies other than MPN
  * Pregnant or lactating women should be excluded due to potential risks associated with cardiovascular evaluations.
  * at age group below 18 years old.
  * who refused to participate in the study.
  Interventions: Other: participants are not assigned an intervention as part of the study
- 40 healthy patients: An external control group will consist of age- and gender-matched individuals without any hematological disorders or significant cardiovascular conditions. They will be recruited from health care workers
  Interventions: Other: participants are not assigned an intervention as part of the study

INTERVENTIONS:
Other: participants are not assigned an intervention as part of the study — participants are not assigned an intervention as part of the study
  Other Names: participants are not assigned an intervention as part of the study.

SUMMARY:
The primary aim of this research is to investigate the clinical and subclinical cardiovascular complications and its relationship with myeloproliferative neoplasms seeking to assess incidence, prevalence and severity in comparison to healthy group and analyze potential risk factors including genetic mutations, inflammatory markers and hematological parameters

DETAILED DESCRIPTION:
Myeloproliferative neoplasms (MPNs) are a group of hematological disorders characterized by clonal proliferation of stem cells leading to excessive production of blood cells. The primary types include polycythemia vera, essential thrombocythemia, and primary myelofibrosis. They share a common characteristic in that they lack the Philadelphia chromosome.

Patients with MPN face an elevated risk of various clinical cardiovascular complications including arterial and venous thromboembolism, hypertension and heart failure. This increased risk can be attributed to several factors including, chronic inflammation, hyperviscosity due to increased blood cells count and genetic mutation like JAK2 V617F which plays a pivotal role in disease pathogenesis.

While clinical cardiovascular events in MPN patients are well-documented, subclinical manifestations such as subclinical atherosclerosis, pulmonary hypertension, left ventriclar hypertrophy, diastolic dysfunction and arrhythmia are often overlooked. These subclinical changes may significantly contribute to morbidity and mortality but are not routinely assessed in clinical practice. Non invasive modalities such as electrocardiography, echocardiography, carotid doppler ultrasound and limb doppler ultrasound can provide vulnerable tools for early detection of these cardiovascular manifestations.

So understanding the relationship between myloproliferative neoplasms and incidence and severity of cardiovascular complications is crucial. This knowledge can enhance risk assessment, improve patient care and outcomes and facilitate targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed diagnosis of myeloproliferative neoplasms of one of the following:
* Essential thrombocythemia (ET)
* Polycythemia vera (PV)
* Primary myelofibrosis (PMF)
* Adults aged 18 years and older.
* who accept to participate in the study in Assiut university hospital.

Exclusion Criteria:

* Patients with secondary erythrocytosis or thrombocytosis due to other underlying conditions (e.g., chronic hypoxia, tumors) will be excluded.
* Patients who have experienced a myocardial infarction, stroke, heart failure, Hypertension, or significant cardiovascular event before diagnosis of MPN
* Patients with severe comorbid conditions that could confound results, such as:
* Severe renal or hepatic impairment
* Active malignancies other than MPN
* Pregnant or lactating women should be excluded due to potential risks associated with cardiovascular evaluations.
* at age group below 18 years old.
* who refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults aged 18-75 years Participants with MPN will be recruited from clinical Haematology Unit of the Internal Medicine at Assiut university while healthy participants will be recruited from health care workers Inclusion criteria of MPN patients will include individuals diagnosed with myeloproliferative neoplasms: essential thrombocythemia, Polycythemia vera and Primary myelofibrosis Exclusion criteria of MPN patients will encompass individuals with secondary erythrocytosis or thrombocytosis due to other underlying conditions (e.g., chronic hypoxia, tumors) , patients who have experienced a myocardial infarction, stroke, heart failure, Hypertension, or significant cardiovascular event before diagnosis of MPN, Patients with severe comorbid conditions that could confound results, such as: Severe renal or hepatic impairment and Active malignancies other than MPN and pregnant and lactating women Study will take place in Assiut university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Cardiovascular Disease and cardiovascular Risk Factors | through study completion, an average of 4 years
  Assessment of clinical cardiovascular disease (CVD) through patient history, physical examination, and diagnostic tests (e.g., ECG, echocardiography) and Measurement of risk factors such as:
  * Blood pressure (systolic and diastolic)
  * Lipid profile (total cholesterol, LDL, HDL, triglycerides)
  * Body mass index (BMI) kg/m^2

SECONDARY OUTCOMES:
Subclinical Cardiovascular Manifestations and Comparison with the healthy control group | through study completion, an average of 4 years
  Subclinical cardiovascular manifestations will be detected by using of imaging techniques such as:
  * Carotid artery doppler ultrasound
  * limb doppler ultrasound

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guglielmelli P, Gangat N, Coltro G, Lasho TL, Loscocco GG, Finke CM, Morsia E, Sordi B, Szuber N, Hanson CA, Pardanani A, Vannucchi AM, Tefferi A. Mutations and thrombosis in essential thrombocythemia. Blood Cancer J. 2021 Apr 27;11(4):77. doi: 10.1038/s41408-021-00470-y. No abstract available. PMID 33907189
- [Background] Leiva O, Bekendam RH, Garcia BD, Thompson C, Cantor A, Chitalia V, Ravid K. Emerging Factors Implicated in Fibrotic Organ-Associated Thrombosis: The Case of Two Organs. TH Open. 2019 Jun 7;3(2):e165-e170. doi: 10.1055/s-0039-1692204. eCollection 2019 Apr. PMID 31259299
- [Background] Hultcrantz M, Wilkes SR, Kristinsson SY, Andersson TM, Derolf AR, Eloranta S, Samuelsson J, Landgren O, Dickman PW, Lambert PC, Bjorkholm M. Risk and Cause of Death in Patients Diagnosed With Myeloproliferative Neoplasms in Sweden Between 1973 and 2005: A Population-Based Study. J Clin Oncol. 2015 Jul 10;33(20):2288-95. doi: 10.1200/JCO.2014.57.6652. Epub 2015 Jun 1. PMID 26033810
- [Background] Tefferi A, Guglielmelli P, Larson DR, Finke C, Wassie EA, Pieri L, Gangat N, Fjerza R, Belachew AA, Lasho TL, Ketterling RP, Hanson CA, Rambaldi A, Finazzi G, Thiele J, Barbui T, Pardanani A, Vannucchi AM. Long-term survival and blast transformation in molecularly annotated essential thrombocythemia, polycythemia vera, and myelofibrosis. Blood. 2014 Oct 16;124(16):2507-13; quiz 2615. doi: 10.1182/blood-2014-05-579136. Epub 2014 Jul 18. PMID 25037629
- [Background] Fidler TP, Xue C, Yalcinkaya M, Hardaway B, Abramowicz S, Xiao T, Liu W, Thomas DG, Hajebrahimi MA, Pircher J, Silvestre-Roig C, Kotini AG, Luchsinger LL, Wei Y, Westerterp M, Snoeck HW, Papapetrou EP, Schulz C, Massberg S, Soehnlein O, Ebert B, Levine RL, Reilly MP, Libby P, Wang N, Tall AR. The AIM2 inflammasome exacerbates atherosclerosis in clonal haematopoiesis. Nature. 2021 Apr;592(7853):296-301. doi: 10.1038/s41586-021-03341-5. Epub 2021 Mar 17. PMID 33731931
- [Background] Garypidou V, Vakalopoulou S, Dimitriadis D, Tziomalos K, Sfikas G, Perifanis V. Incidence of pulmonary hypertension in patients with chronic myeloproliferative disorders. Haematologica. 2004 Feb;89(2):245-6. No abstract available. PMID 15003906
- [Background] Briukhovetska D, Dorr J, Endres S, Libby P, Dinarello CA, Kobold S. Interleukins in cancer: from biology to therapy. Nat Rev Cancer. 2021 Aug;21(8):481-499. doi: 10.1038/s41568-021-00363-z. Epub 2021 Jun 3. PMID 34083781